CLINICAL TRIAL: NCT04553471
Title: A Trial of Palliative Lattice Stereotactic Body Radiotherapy (SBRT) for Patients With Sarcoma, Thoracic, Abdominal, and Pelvic Cancers
Brief Title: Palliative Lattice Stereotactic Body Radiotherapy (SBRT) for Patients With Sarcoma, Thoracic, Abdominal, and Pelvic Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Goldman Sachs Foundation (Emerson Collective) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202009022
Record Dates: First submitted 2020-09-09; First posted 2020-09-17 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Sarcoma; Thoracic Cancer; Abdominal Cancer; Pelvic Cancer
MeSH Terms: conditions — Sarcoma; Pelvic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: At least 10 participants will be enrolled in each cohort (soft tissue sarcomas, thoracic cancers, abdominal, and pelvic cancers).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SBRT (Experimental): 5-fraction Lattice SBRT delivered to 20 Gy with a simultaneous integrated boost (SIB) to 66.7 Gy.
  Interventions: Radiation: Stereotactic body radiotherapy; Procedure: Research blood draw

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Treatment will take approximately 2 weeks.
  Other Names: SBRT
Procedure: Research blood draw — -Baseline, immediately after radiotherapy completion (fraction 5), 14 days after radiotherapy, and 30 day follow-up

SUMMARY:
This is a study evaluating the safety and efficacy of Lattice SBRT for patients with large tumors (≥ 4.5 cm) planning to undergo palliative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed sarcoma (including extremity), thoracic cancer (including esophageal), abdominal cancer (including retroperitoneal sarcoma), or pelvic cancer.
* Planning to undergo palliative radiotherapy to a lesion ≥ 4.5 cm as measured with radiographic imaging or with calipers by clinical exam.
* ECOG performance status ≤ 2
* At least 18 years of age.
* Radiotherapy is known to be teratogenic. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 6 months after completion of the study
* Ability to understand and willingness to sign an IRB approved written informed consent document

Exclusion Criteria:

* Prior high-dose radiotherapy that overlaps with any planned site of protocol radiotherapy. Patients where the Lattice SBRT fields may overlap with the low dose (<10 Gy) region of prior radiotherapy treatments are eligible and may be treated if this is determined to be safe by the treating physician.
* Patients with tumors in need of urgent surgical intervention, such as life-threatening bleeding or those at high risk for pathologic fracture.
* Currently receiving any cytotoxic cancer therapy regimens or VEGF inhibitors that will overlap with the Lattice SBRT administration.

  *Cytotoxic chemotherapy and VEGF inhibitors prior to radiotherapy or planned after radiotherapy delivery are allowed at the discretion of the treating radiation oncologist. This includes continuing a treatment plan which was initiated prior to the start of radiotherapy. A 2-week washout is recommended, but not required.
* Pregnant. Women of childbearing potential must have a negative pregnancy test within 20 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended. Recommend exclusion of specific ART agents based on predicted drug-drug interactions (i.e. for sensitive CYP3A4 substrates, concurrent strong CYP3A4 inhibitors (ritonavir and cobicistat) or inducers (efavirenz) should be contraindicated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Samson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duriseti S, Kavanaugh J, Goddu S, Price A, Knutson N, Reynoso F, Michalski J, Mutic S, Robinson C, Spraker MB. Spatially fractionated stereotactic body radiation therapy (Lattice) for large tumors. Adv Radiat Oncol. 2021 Jan 8;6(3):100639. doi: 10.1016/j.adro.2020.100639. eCollection 2021 May-Jun. PMID 34195486
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SBRT
Started | 70
Completed | 66
Not Completed | 4
Not completed — Did not start treatment on protocol | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | SBRT
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 65.5 [19 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 69
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 57
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Rate of Local Control
Time Frame: At 6 months
Population: Participants must have received treatment and had a 6 month disease assessment to be evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT
Number analyzed (Participants) | 32
Participants | 29

2. Primary Outcome: Number of Participants With Treatment-related, Non-hematologic Grade ≥ 3 Toxicity
Description: -Graded using CTCAE v5.0
Time Frame: Through 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT
Number analyzed (Participants) | 66
Participants | 2

3. Secondary Outcome: Mean Change From Baseline - PROMIS Physical Function Assessment
Description: * Each value is the mean of the changes from baseline PROMIS T-Score to timepoint PROMIS T-score.
  * PROMIS Physical Function is a 10-item questionnaire assessing current self-reported physical function with answers ranging from 1 = cannot do to 5 = not at all/without any difficulty.
  * A PROMIS T-Score of 50 corresponds to the mean of the general population. A magnitude of 10 on the PROMIS scale corresponds to a standard deviation.
  * A high T-Score for PROMIS Physical Function Assessment correlates to a higher physical function, or positive outcome. Since the scale is standardized a score of 60 is one standard deviation higher, or better functioning, than the reference population mean.
Time Frame: 2 weeks post-treatment (approximately week 4), 30 days, 3 months, 6 months, and 12 months
Population: If a participant did not complete the questionnaire at the timepoint then they are not included.
Measure: Mean (Standard Deviation); unit: T-Score
Groups:
- SBRT-2 Weeks Post Treatment; SBRT-30 Days; SBRT-3 Months; SBRT-6 Months; SBRT-12 Months: 5-fraction Lattice SBRT delivered to 20 Gy with a simultaneous integrated boost (SIB) to 66.7 Gy.
Arm/Group | SBRT-2 Weeks Post Treatment | SBRT-30 Days | SBRT-3 Months | SBRT-6 Months | SBRT-12 Months
Number analyzed (Participants) | 38 | 39 | 31 | 21 | 15
T-Score | 2.22 (5.976098077) | -0.27 (6.464353622) | 2.01 (8.493109161) | 2.76 (8.144051291) | -0.72 (6.097212478)

4. Secondary Outcome: Mean Change From Baseline-PROMIS Global Health Physical Assessment
Description: * Each value is the mean of the changes from baseline PROMIS T-Score to timepoint PROMIS T-score.
  * PROMIS Global Health is a 2-item questionnaire assessing current self-reported physical function with answers ranging from 1=poor/not all all to 5=excellent/completely
  * A PROMIS T-Score of 50 corresponds to the mean of the general population. A magnitude of 10 on the PROMIS scale corresponds to a standard deviation.
  * A high T-Score for PROMIS Global Health Physical Assessment correlates to a higher global health physical assessment, or positive outcome. Since the scale is standardized a score of 60 is one standard deviation higher, or better physical assessment, than the reference population mean
Time Frame: 2 weeks post-treatment (approximately week 4), 30 days, 3 months, 6 months, and 12 months
Population: If a participant did not complete the questionnaire at the timepoint then they are not included.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | SBRT-2 Weeks Post Treatment | SBRT-30 Days | SBRT-3 Months | SBRT-6 Months | SBRT-12 Months
Number analyzed (Participants) | 41 | 39 | 31 | 20 | 16
T-Score | 1.36 (4.885644726) | 0.40 (5.629643682) | 0.95 (6.704716684) | 2.63 (7.152040563) | 1.06 (5.996095952)

5. Secondary Outcome: Mean Change From Baseline-PROMIS Depression Assessment
Description: * Each value is the mean of the changes from baseline PROMIS T-Score to timepoint PROMIS T-score.
  * PROMIS Depression is a 4-item questionnaire assessing current self-reported depression with answers ranging from 1=never to 5=always
  * A PROMIS T-Score of 50 corresponds to the mean of the general population. A magnitude of 10 on the PROMIS scale corresponds to a standard deviation.
  * A high T-Score for PROMIS Depression Assessment correlates to more depression, or negative outcome. Since the scale is standardized a score of 60 is one standard deviation higher, or worse depression, than the reference population mean
Time Frame: 2 weeks post-treatment (approximately week 4), 30 days, 3 months, 6 months, and 12 months
Population: If a participant did not complete the questionnaire at the timepoint then they are not included.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | SBRT-2 Weeks Post Treatment | SBRT-30 Days | SBRT-3 Months | SBRT-6 Months | SBRT-12 Months
Number analyzed (Participants) | 40 | 39 | 32 | 20 | 16
T-Score | 1.01 (6.575515969) | 0.72 (7.013388007) | -0.15 (7.290691563) | 1.01 (9.929482946) | -2.43 (8.78069853)

6. Secondary Outcome: Mean Change From Baseline-PROMIS Anxiety Assessment
Description: * Each value is the mean of the changes from baseline PROMIS T-Score to timepoint PROMIS T-score.
  * PROMIS Anxiety is a 29-item questionnaire assessing current self-reported anxiety with answers ranging from 1=never to 5=always
  * A PROMIS T-Score of 50 corresponds to the mean of the general population. A magnitude of 10 on the PROMIS scale corresponds to a standard deviation.
  * A high T-Score for PROMIS Anxiety Assessment correlates to more anxiety, or negative outcome. Since the scale is standardized a score of 60 is one standard deviation higher, or worse anxiety, than the reference population mean.
Time Frame: 2 weeks post-treatment (approximately week 4), 30 days, 3 months, 6 months, and 12 months
Population: If a participant did not complete the questionnaire at the timepoint then they are not included.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | SBRT-2 Weeks Post Treatment | SBRT-30 Days | SBRT-3 Months | SBRT-6 Months | SBRT-12 Months
Number analyzed (Participants) | 42 | 40 | 32 | 20 | 16
T-Score | 1.16 (7.520188855) | 0.12 (6.799064792) | -1.66 (8.797717813) | -0.15 (8.436791296) | -4.34 (9.955565864)

7. Secondary Outcome: Mean Change From Baseline-Numeric Pain Scale
Description: * Each value is the mean of the changes from baseline Numeric Pain Scale score to timepoint Numeric Pain Scale score.
  * The Numeric Pain Scale is an 11-point scale for patient self-reporting of pain
  * The Numeric Pain Rating Scale (NPRS) measures pain intensity in adults using a scale from 0 or "no pain" to 10 or "worst possible pain." This measure is unidimensional and evaluated on the 0-10 scale. A higher value on the scale correlates with a worse pain and a worse outcome.
Time Frame: 2 weeks post-treatment (approximately week 4), 30 days, 3 months, 6 months, and 12 months
Population: If a participant did not complete the questionnaire at the timepoint then they are not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SBRT-2 Weeks Post Treatment | SBRT-30 Days | SBRT-3 Months | SBRT-6 Months | SBRT-12 Months
Number analyzed (Participants) | 23 | 24 | 18 | 14 | 13
score on a scale | 0.87 (3.911571967) | -0.38 (4.209848701) | -0.83 (2.357715744) | -0.29 (3.709210396) | -0.77 (2.832956234)

8. Secondary Outcome: Patient Reported Toxicity as Measured by PRO-CTCAE Assessment (Gastrointestinal Cancer Sites)
Description: * The PRO-CTCAE Measurement System characterizes the frequency, severity, interference, and presence/absence of symptomatic toxicities. The higher the score the worst the symptoms.
  * Severity options include none=1, mild=2, moderate=3, severe = 4, very severe=5.
  * Interference options include not at all=1, a little bit=2, somewhat=3, quite a bit=4, very much=5
  * Frequency options include never=1, rarely=2, occasionally=3, frequently=4, almost constantly=5
Time Frame: Baseline, 2 weeks post-treatment (approximately week 4), 30 days, 3 months, 6 months, and 12 months
Population: If a participant did not complete the questionnaire at the timepoint then they are not included. If the participant did not answer a question on the questionnaire then they are not included for that question.
Measure: Median (Full Range); unit: score on a scale
Groups:
- SBRT - Baseline; SBRT - 2 Weeks Post-treatment; SBRT - 30 Days; SBRT - 3 Months; SBRT - 6 Months; SBRT - 12 Months: 5-fraction Lattice SBRT delivered to 20 Gy with a simultaneous integrated boost (SIB) to 66.7 Gy.
Arm/Group | SBRT - Baseline | SBRT - 2 Weeks Post-treatment | SBRT - 30 Days | SBRT - 3 Months | SBRT - 6 Months | SBRT - 12 Months
Number analyzed (Participants) | 20 | 15 | 15 | 12 | 9 | 5
score on a scale
  Severity of decreased appetite: number analyzed (Participants) | 20 | 15 | 15 | 12 | 8 | 5
  Severity of decreased appetite | 2 [1 to 5] | 3 [1 to 5] | 2 [1 to 5] | 2 [1 to 4] | 3 [1 to 3] | 1 [1 to 3]
  Decreased appetite interference: number analyzed (Participants) | 20 | 15 | 15 | 11 | 8 | 5
  Decreased appetite interference | 1 [1 to 4] | 3 [1 to 5] | 1 [1 to 5] | 1 [1 to 3] | 1 [1 to 5] | 1 [1 to 3]
  Frequency of nausea: number analyzed (Participants) | 20 | 15 | 15 | 12 | 8 | 5
  Frequency of nausea | 1 [1 to 5] | 2 [1 to 5] | 2 [1 to 5] | 1 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
  Severity of nausea: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Severity of nausea | 1 [1 to 5] | 2 [1 to 4] | 2 [1 to 5] | 1 [1 to 2] | 2 [1 to 2] | 2 [1 to 3]
  Frequency of vomiting: number analyzed (Participants) | 20 | 15 | 15 | 12 | 8 | 5
  Frequency of vomiting | 1 [1 to 5] | 1 [1 to 3] | 1 [1 to 5] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3]
  Severity of vomiting: number analyzed (Participants) | 20 | 14 | 15 | 11 | 8 | 5
  Severity of vomiting | 1 [1 to 4] | 1 [1 to 2] | 1 [1 to 5] | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 3]
  Frequency of heartburn: number analyzed (Participants) | 20 | 15 | 15 | 12 | 8 | 5
  Frequency of heartburn | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3]
  Severity of heartburn: number analyzed (Participants) | 20 | 14 | 14 | 11 | 8 | 5
  Severity of heartburn | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3]
  Frequency of bloating: number analyzed (Participants) | 20 | 15 | 15 | 12 | 8 | 5
  Frequency of bloating | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 5] | 1.5 [1 to 4] | 2 [1 to 4] | 1 [1 to 3]
  Severity of bloating: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Severity of bloating | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 5] | 1 [1 to 3] | 2 [1 to 5] | 1 [1 to 2]
  Frequency of hiccups: number analyzed (Participants) | 20 | 15 | 15 | 12 | 8 | 5
  Frequency of hiccups | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 5] | 1 [1 to 2]
  Severity of hiccups: number analyzed (Participants) | 19 | 15 | 14 | 12 | 8 | 5
  Severity of hiccups | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 4] | 1 [1 to 2]
  Severity of constipation: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Severity of constipation | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 4] | 1 [1 to 2] | 2 [1 to 3] | 1 [1 to 1]
  Frequency of diarrhea: number analyzed (Participants) | 19 | 14 | 15 | 12 | 8 | 5
  Frequency of diarrhea | 1 [1 to 4] | 1.5 [1 to 5] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2]
  Frequency of abdominal pain: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Frequency of abdominal pain | 2 [1 to 5] | 3 [1 to 5] | 3 [1 to 5] | 2 [1 to 4] | 3 [1 to 5] | 2 [1 to 4]
  Severity of abdominal pain: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Severity of abdominal pain | 2 [1 to 5] | 2.5 [1 to 5] | 2 [1 to 5] | 2 [1 to 3] | 2 [1 to 4] | 2 [1 to 3]
  Abdominal pain interference: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Abdominal pain interference | 1 [1 to 5] | 2 [1 to 5] | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3]
  Frequency of bowel movement control loss: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Frequency of bowel movement control loss | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
  Bowel movement control loss interference: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Bowel movement control loss interference | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 1] | 1 [1 to 2] | 1 [1 to 4] | 1 [1 to 2]
  Severity of numbness/tingling in hands or feet: number analyzed (Participants) | 19 | 14 | 15 | 12 | 8 | 5
  Severity of numbness/tingling in hands or feet | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 2]
  Numbness or tingling in hands or feet interference: number analyzed (Participants) | 20 | 13 | 14 | 11 | 8 | 5
  Numbness or tingling in hands or feet interference | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2]
  Severity of dizziness: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Severity of dizziness | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 3]
  Dizziness interference: number analyzed (Participants) | 20 | 13 | 14 | 10 | 7 | 5
  Dizziness interference | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
  Severity of concentration problems: number analyzed (Participants) | 20 | 14 | 15 | 12 | 8 | 5
  Severity of concentration problems | 1 [1 to 4] | 1.5 [1 to 4] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2]
  Concentration problems interference: number analyzed (Participants) | 20 | 14 | 15 | 11 | 8 | 5
  Concentration problems interference | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
  Severity of memory problems: number analyzed (Participants) | 20 | 14 | 15 | 11 | 8 | 5
  Severity of memory problems | 1 [1 to 3] | 2 [1 to 4] | 2 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2]
  Memory problem interference: number analyzed (Participants) | 20 | 13 | 14 | 12 | 8 | 5
  Memory problem interference | 1 [1 to 3] | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
  Frequency of pain: number analyzed (Participants) | 20 | 15 | 14 | 12 | 9 | 5
  Frequency of pain | 3 [1 to 5] | 4 [1 to 5] | 4 [2 to 5] | 3 [1 to 4] | 2 [1 to 5] | 2 [1 to 4]
  Severity of pain: number analyzed (Participants) | 20 | 15 | 15 | 11 | 9 | 5
  Severity of pain | 3 [1 to 5] | 3 [1 to 5] | 3 [1 to 5] | 2 [1 to 4] | 2 [1 to 5] | 2 [1 to 3]
  Pain interference: number analyzed (Participants) | 20 | 15 | 15 | 11 | 9 | 5
  Pain interference | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 5] | 1 [1 to 2] | 2 [1 to 5] | 1 [1 to 2]
  Severity of insomnia: number analyzed (Participants) | 20 | 15 | 15 | 12 | 9 | 4
  Severity of insomnia | 2 [1 to 5] | 3 [1 to 5] | 2 [1 to 5] | 1.5 [1 to 4] | 2 [1 to 5] | 1 [1 to 4]
  Insomnia interference | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 4] | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 4]
  Severity of fatigue | 3 [1 to 5] | 3 [2 to 5] | 3 [1 to 5] | 3 [1 to 4] | 3 [1 to 4] | 2 [2 to 4]
  Fatigue interference | 3 [1 to 5] | 3 [1 to 5] | 3 [1 to 5] | 2.5 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]
  Frequency of anxiety: number analyzed (Participants) | 20 | 14 | 15 | 12 | 9 | 5
  Frequency of anxiety | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 2 [1 to 4]
  Severity of anxiety | 2 [1 to 4] | 1 [1 to 3] | 2 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 2 [1 to 3]
  Anxiety interference: number analyzed (Participants) | 20 | 13 | 15 | 12 | 9 | 5
  Anxiety interference | 1 [1 to 5] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 4]
  Frequency of depression | 1 [1 to 5] | 1 [1 to 5] | 2 [1 to 3] | 1 [1 to 3] | 1 [1 to 5] | 1 [1 to 4]
  Severity of depression: number analyzed (Participants) | 19 | 15 | 15 | 12 | 9 | 5
  Severity of depression | 1 [1 to 5] | 1 [1 to 5] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 5] | 1 [1 to 4]
  Depression interference: number analyzed (Participants) | 19 | 14 | 15 | 12 | 9 | 5
  Depression interference | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 5] | 1 [1 to 4]
  Frequency of sadness or unhappiness | 2 [1 to 4] | 2 [1 to 5] | 2 [1 to 5] | 1.5 [1 to 3] | 2 [1 to 4] | 1 [1 to 4]
  Severity of sadness or unhappiness: number analyzed (Participants) | 19 | 15 | 15 | 12 | 9 | 5
  Severity of sadness or unhappiness | 2 [1 to 4] | 2 [1 to 5] | 2 [1 to 3] | 1 [1 to 3] | 2 [1 to 4] | 1 [1 to 4]
  Sadness or happiness interference | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 3]

9. Secondary Outcome: Patient Reported Toxicity as Measured by PRO-CTCAE Assessment (Pelvic Cancer Sites)
Description: * The PRO-CTCAE Measurement System characterizes the frequency, severity, interference, and presence/absence of symptomatic toxicities. The higher the score the worst the symptoms.
  * Severity options include none=1, mild=2, moderate=3, severe = 4, very severe=5.
  * Interference options include not at all=1, a little bit=2, somewhat=3, quite a bit=4, very much=5
  * How often options include 1=never, 2=rarely, 3=occasionally, 4=frequently, 5=almost constantly
  * Severity of difficulty getting/keeping erection, ejaculation problems, decreased sexual interest, vaginal pain 1=none, 2=mild, 3=moderate, 4=severe, 5=very severe
  * Experienced unusual vaginal discharge options include 1=not at all, 2=a little bit, 3 = somewhat, 4=quite a bit, 5=very much
Time Frame: Baseline, 2 weeks post-treatment (approximately week 4), 30 days, 3 months, 6 months, and 12 months
Population: as for outcome 8
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SBRT - Baseline | SBRT - 2 Weeks Post-treatment | SBRT - 30 Days | SBRT - 3 Months | SBRT - 6 Months | SBRT - 12 Months
Number analyzed (Participants) | 21 | 14 | 13 | 10 | 7 | 6
score on a scale
  Severity of numbness/tingling in hands or feet: number analyzed (Participants) | 21 | 14 | 12 | 10 | 7 | 6
  Severity of numbness/tingling in hands or feet | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 5] | 2 [1 to 3] | 1.5 [1 to 4]
  Numbness or tingling in hands or feet interference: number analyzed (Participants) | 20 | 12 | 9 | 10 | 6 | 5
  Numbness or tingling in hands or feet interference | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 5] | 1 [1 to 3] | 1 [1 to 4]
  Severity of dizziness: number analyzed (Participants) | 21 | 14 | 12 | 10 | 7 | 6
  Severity of dizziness | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 2 [1 to 2] | 2.5 [1 to 3]
  Dizziness interference: number analyzed (Participants) | 20 | 12 | 9 | 10 | 6 | 5
  Dizziness interference | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 2 [1 to 3]
  Severity of concentration problems: number analyzed (Participants) | 21 | 14 | 12 | 10 | 7 | 6
  Severity of concentration problems | 1 [1 to 4] | 2 [1 to 4] | 1.5 [1 to 5] | 1.5 [1 to 2] | 1 [1 to 2] | 1.5 [1 to 5]
  Concentration problems interference: number analyzed (Participants) | 21 | 13 | 10 | 10 | 6 | 6
  Concentration problems interference | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 2] | 1 [1 to 2] | 1.5 [1 to 5]
  Severity of memory problems: number analyzed (Participants) | 21 | 14 | 12 | 10 | 7 | 6
  Severity of memory problems | 1 [1 to 3] | 2 [1 to 5] | 1 [1 to 5] | 2 [1 to 2] | 1 [1 to 2] | 1.5 [1 to 5]
  Memory problem interference: number analyzed (Participants) | 21 | 13 | 10 | 10 | 7 | 6
  Memory problem interference | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 5] | 1 [1 to 2] | 1 [1 to 1] | 1.5 [1 to 5]
  Frequency of pain: number analyzed (Participants) | 21 | 14 | 13 | 10 | 7 | 5
  Frequency of pain | 4 [1 to 5] | 3.5 [2 to 5] | 3 [1 to 5] | 3.5 [3 to 5] | 3 [2 to 5] | 4 [3 to 4]
  Severity of pain: number analyzed (Participants) | 20 | 14 | 12 | 10 | 7 | 6
  Severity of pain | 3 [1 to 5] | 3 [2 to 5] | 3 [1 to 4] | 3 [2 to 4] | 3 [2 to 5] | 3 [2 to 4]
  Pain interference: number analyzed (Participants) | 21 | 13 | 12 | 10 | 7 | 6
  Pain interference | 3 [1 to 5] | 3 [1 to 5] | 2 [1 to 5] | 3 [1 to 5] | 2 [1 to 5] | 2.5 [2 to 5]
  Severity of insomnia: number analyzed (Participants) | 20 | 14 | 13 | 10 | 7 | 6
  Severity of insomnia | 2 [1 to 4] | 2 [1 to 3] | 2 [1 to 5] | 1 [1 to 4] | 3 [1 to 5] | 3 [1 to 4]
  Insomnia interference: number analyzed (Participants) | 21 | 14 | 11 | 10 | 6 | 6
  Insomnia interference | 1 [1 to 4] | 1 [1 to 3] | 2 [1 to 5] | 1 [1 to 5] | 3 [1 to 5] | 2.5 [1 to 5]
  Severity of fatigue | 3 [1 to 5] | 3 [2 to 5] | 1 [1 to 5] | 3.5 [1 to 5] | 3 [1 to 4] | 3 [2 to 5]
  Fatigue interference | 3 [1 to 5] | 3 [1 to 5] | 2 [1 to 5] | 3.5 [1 to 5] | 3 [1 to 4] | 2.5 [2 to 5]
  Frequency of anxiety: number analyzed (Participants) | 21 | 13 | 13 | 10 | 7 | 6
  Frequency of anxiety | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 3] | 3 [2 to 5]
  Severity of anxiety: number analyzed (Participants) | 21 | 13 | 11 | 10 | 7 | 6
  Severity of anxiety | 2 [1 to 4] | 2 [1 to 3] | 2 [1 to 5] | 2 [1 to 4] | 2 [1 to 3] | 2.5 [2 to 4]
  Anxiety interference: number analyzed (Participants) | 21 | 13 | 11 | 10 | 7 | 6
  Anxiety interference | 1 [1 to 4] | 2 [1 to 4] | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 3] | 2 [1 to 5]
  Frequency of depression: number analyzed (Participants) | 21 | 14 | 13 | 9 | 7 | 6
  Frequency of depression | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 3] | 1.5 [1 to 4]
  Severity of depression: number analyzed (Participants) | 21 | 14 | 12 | 9 | 7 | 6
  Severity of depression | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 5] | 1 [1 to 3] | 1 [1 to 3] | 1.5 [1 to 4]
  Depression interference: number analyzed (Participants) | 21 | 14 | 12 | 9 | 6 | 6
  Depression interference | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 1] | 1.5 [1 to 4]
  Frequency of sadness or unhappiness: number analyzed (Participants) | 21 | 14 | 13 | 9 | 7 | 6
  Frequency of sadness or unhappiness | 2 [1 to 4] | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 3] | 2 [1 to 4] | 2 [1 to 3]
  Severity of sadness or unhappiness: number analyzed (Participants) | 21 | 13 | 11 | 9 | 7 | 6
  Severity of sadness or unhappiness | 2 [1 to 4] | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 3] | 2 [1 to 4] | 2 [1 to 4]
  Sadness or happiness interference: number analyzed (Participants) | 21 | 13 | 11 | 9 | 6 | 6
  Sadness or happiness interference | 1 [1 to 5] | 1 [1 to 5] | 1 [1 to 5] | 1 [1 to 3] | 1 [1 to 3] | 1.5 [1 to 3]
  Experienced unusual vaginal discharge: number analyzed (Participants) | 14 | 8 | 7 | 8 | 4 | 5
  Experienced unusual vaginal discharge | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 3] | 1 [1 to 1] | 1 [1 to 1]
  Severity of vaginal dryness: number analyzed (Participants) | 14 | 7 | 7 | 7 | 4 | 5
  Severity of vaginal dryness | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 4] | 1 [1 to 1] | 1 [1 to 4] | 1 [1 to 1]
  Severity of pain/burning with urination: number analyzed (Participants) | 17 | 13 | 11 | 9 | 7 | 5
  Severity of pain/burning with urination | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 1] | 1 [1 to 2]
  Frequency of urge to urinate: number analyzed (Participants) | 20 | 14 | 13 | 10 | 7 | 6
  Frequency of urge to urinate | 1.5 [1 to 4] | 2 [1 to 4] | 2 [1 to 4] | 1.5 [1 to 4] | 1 [1 to 4] | 2.5 [1 to 4]
  Urge to urinate interference: number analyzed (Participants) | 21 | 14 | 12 | 10 | 7 | 6
  Urge to urinate interference | 1 [1 to 4] | 1 [1 to 5] | 1.5 [1 to 5] | 1 [1 to 4] | 1 [1 to 2] | 2 [1 to 4]
  Frequency of urination frequency: number analyzed (Participants) | 20 | 14 | 13 | 9 | 7 | 6
  Frequency of urination frequency | 1 [1 to 4] | 2 [1 to 4] | 2 [1 to 5] | 2 [1 to 4] | 1 [1 to 4] | 2.5 [1 to 3]
  Frequent urination interfering: number analyzed (Participants) | 20 | 13 | 12 | 9 | 7 | 6
  Frequent urination interfering | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 3] | 1.5 [1 to 4]
  Frequency of urine leakage: number analyzed (Participants) | 21 | 14 | 13 | 9 | 7 | 6
  Frequency of urine leakage | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 4]
  Urine leakage frequency: number analyzed (Participants) | 20 | 14 | 12 | 9 | 6 | 6
  Urine leakage frequency | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 5] | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 4]
  Severity of difficulty getting/keeping an erection: number analyzed (Participants) | 9 | 3 | 4 | 3 | 2 | 3
  Severity of difficulty getting/keeping an erection | 1 [1 to 5] | 3 [1 to 4] | 2 [1 to 4] | 1 [1 to 3] | 2.5 [1 to 4] | 1 [1 to 5]
  Frequency of ejaculation problems: number analyzed (Participants) | 8 | 2 | 4 | 3 | 2 | 3
  Frequency of ejaculation problems | 1 [1 to 4] | 2 [1 to 3] | 2 [1 to 4] | 1 [1 to 3] | 2.5 [1 to 4] | 1 [1 to 5]
  Severity of decreased sexual interest: number analyzed (Participants) | 10 | 4 | 6 | 5 | 3 | 4
  Severity of decreased sexual interest | 1.5 [1 to 5] | 2 [1 to 4] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 5] | 1 [1 to 5]
  Severity of pain during vaginal sex: number analyzed (Participants) | 5 | 0 | 1 | 3 | 2 | 3
  Severity of pain during vaginal sex | 1 [1 to 1] |  | 1 [NA to NA] — Only 1 participant was evaluable. | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]

10. Secondary Outcome: Patient Reported Toxicity as Measured by PRO-CTCAE Assessment (Sarcoma Cancer Sites)
Description: as for outcome 8
Time Frame: Baseline, 2 weeks post-treatment (approximately week 4), 30 days, 3 months, 6 months, and 12 months
Population: as for outcome 8
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SBRT - Baseline | SBRT - 2 Weeks Post-treatment | SBRT - 30 Days | SBRT - 3 Months | SBRT - 6 Months | SBRT - 12 Months
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 1 | 0
score on a scale
  Severity of dry mouth | 1.5 [1 to 2] | 1 [1 to 5] | 1 [1 to 1] | 2 [1 to 3] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of difficulty swallowing | 2 [1 to 3] | 2 [1 to 4] | 1.5 [1 to 2] | 1.5 [1 to 2] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of mouth or throat sores | 1 [1 to 1] | 1 [1 to 4] | 2 [1 to 3] | 1 [1 to 1] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Mouth or throat sores interference | 1 [1 to 1] | 1 [1 to 1] | 1.5 [1 to 2] | 1 [1 to 1] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of skin cracking at corners of mouth | 1 [1 to 1] | 3 [1 to 4] | 1 [1 to 1] | 1.5 [1 to 2] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of hoarse voice | 1.5 [1 to 2] | 3 [1 to 3] | 1 [1 to 1] | 1 [1 to 1] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of numbness/tingling in hands or feet | 3 [2 to 4] | 1 [1 to 5] | 2.5 [1 to 4] | 3.5 [3 to 4] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Numbness or tingling in hands or feet interference | 2 [1 to 3] | 1 [1 to 5] | 2 [1 to 3] | 2 [1 to 3] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of dizziness | 3 [1 to 5] | 1 [1 to 3] | 2 [2 to 2] | 1 [1 to 1] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Dizziness interference | 2.5 [1 to 4] | 1 [1 to 3] | 2 [2 to 2] | 1 [1 to 1] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of concentration problems | 1 [1 to 1] | 1 [1 to 2] | 1.5 [1 to 2] | 1 [1 to 1] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Concentration problems interference | 1 [1 to 1] | 1 [1 to 2] | 1.5 [1 to 2] | 1 [1 to 1] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of memory problems | 1 [1 to 1] | 1 [1 to 2] | 1.5 [1 to 2] | 1 [1 to 1] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Memory problem interference | 1 [1 to 1] | 1 [1 to 3] | 1.5 [1 to 2] | 1 [1 to 1] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Frequency of pain | 3 [2 to 4] | 4 [4 to 4] | 4.5 [4 to 5] | 4.5 [4 to 5] | 2 [NA to NA] — Only 1 participant was evaluable. |
  Severity of pain | 2.5 [2 to 3] | 4 [4 to 5] | 4.5 [4 to 5] | 4 [4 to 4] | 2 [NA to NA] — Only 1 participant was evaluable. |
  Pain interference | 2.5 [1 to 4] | 3 [3 to 3] | 4 [3 to 5] | 3 [3 to 3] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of insomnia: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Severity of insomnia | 2 [1 to 3] | 3 [1 to 5] | 3 [3 to 3] | 1.5 [1 to 2] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Insomnia interference: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Insomnia interference | 2 [1 to 3] | 2.5 [1 to 4] | 3 [2 to 4] | 1.5 [1 to 2] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of fatigue: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Severity of fatigue | 3.5 [2 to 5] | 3.5 [2 to 5] | 2 [2 to 2] | 2 [1 to 3] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Fatigue interference: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Fatigue interference | 3.5 [2 to 5] | 3.5 [2 to 5] | 2 [2 to 2] | 1.5 [1 to 2] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Frequency of anxiety: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Frequency of anxiety | 2 [1 to 3] | 2.5 [1 to 4] | 1.5 [1 to 2] | 2 [1 to 3] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Severity of anxiety: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Severity of anxiety | 2 [1 to 3] | 2.5 [1 to 4] | 1.5 [1 to 2] | 2 [1 to 3] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Anxiety interference: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Anxiety interference | 2 [1 to 3] | 2 [1 to 3] | 1 [1 to 1] | 2 [1 to 3] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Frequency of depression: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Frequency of depression | 1.5 [1 to 2] | 2 [1 to 3] | 1 [1 to 1] | 1.5 [1 to 2] | 2 [NA to NA] — Only 1 participant was evaluable. |
  Severity of depression: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Severity of depression | 1.5 [1 to 2] | 2 [1 to 3] | 1 [1 to 1] | 2 [1 to 3] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Depression interference: number analyzed (Participants) | 2 | 2 | 2 | 2 | 1 | 0
  Depression interference | 1.5 [1 to 2] | 2 [1 to 3] | 1 [1 to 1] | 2 [1 to 3] | 1 [NA to NA] — Only 1 participant was evaluable. |
  Frequency of sadness or unhappiness | 3 [3 to 3] | 2 [1 to 4] | 2 [2 to 2] | 2.5 [2 to 3] | 2 [NA to NA] — Only 1 participant was evaluable. |
  Severity of sadness or unhappiness | 3.5 [3 to 4] | 2 [1 to 4] | 1.5 [1 to 2] | 2.5 [2 to 3] | 2 [NA to NA] — Only 1 participant was evaluable. |
  Sadness or happiness interference | 2.5 [2 to 3] | 1 [1 to 4] | 1 [1 to 1] | 2 [2 to 2] | 1 [NA to NA] — Only 1 participant was evaluable. |

11. Secondary Outcome: Patient Reported Toxicity as Measured by PRO-CTCAE Assessment (Thoracic Cancer Sites)
Description: as for outcome 8
Time Frame: Baseline, 2 weeks post-treatment (approximately week 4), 30 days, 3 months, 6 months, and 12 months
Population: If a participant did not complete the questionnaire at the timepoint then they are not included.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SBRT - Baseline | SBRT - 2 Weeks Post-treatment | SBRT - 30 Days | SBRT - 3 Months | SBRT - 6 Months | SBRT - 12 Months
Number analyzed (Participants) | 18 | 11 | 11 | 10 | 7 | 5
score on a scale
  Severity of hoarse voice | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1.5 [1 to 3] | 1 [1 to 3] | 1 [1 to 2]
  Severity of decreased appetite | 2 [1 to 4] | 3 [1 to 4] | 2 [1 to 4] | 1.5 [1 to 3] | 1 [1 to 3] | 1 [1 to 3]
  Decreased appetite interference: number analyzed (Participants) | 18 | 11 | 11 | 10 | 6 | 5
  Decreased appetite interference | 1 [1 to 4] | 2 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2]
  Frequency of nausea | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
  Severity of nausea: number analyzed (Participants) | 17 | 10 | 11 | 10 | 6 | 5
  Severity of nausea | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
  Frequency of vomiting | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 3]
  Severity of vomiting: number analyzed (Participants) | 16 | 11 | 11 | 10 | 6 | 5
  Severity of vomiting | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 4] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 3]
  Frequency of heartburn | 1 [1 to 4] | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 3]
  Severity of heartburn: number analyzed (Participants) | 16 | 11 | 11 | 10 | 6 | 5
  Severity of heartburn | 1 [1 to 3] | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 3]
  Frequency of bloating | 1 [1 to 3] | 2 [1 to 4] | 1 [1 to 3] | 2 [1 to 3] | 2 [1 to 3] | 1 [1 to 2]
  Severity of bloating: number analyzed (Participants) | 17 | 11 | 11 | 9 | 7 | 5
  Severity of bloating | 2 [1 to 3] | 2 [1 to 4] | 1 [1 to 4] | 2 [1 to 2] | 2 [1 to 2] | 1 [1 to 2]
  Frequency of hiccups | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 1]
  Severity of hiccups: number analyzed (Participants) | 17 | 10 | 11 | 9 | 7 | 5
  Severity of hiccups | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 1]
  Severity of shortness of breath | 3 [2 to 4] | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 4] | 3 [1 to 3] | 2 [1 to 3]
  Shortness of breath interference | 3 [1 to 5] | 3 [1 to 4] | 2 [1 to 4] | 2 [1 to 4] | 3 [1 to 4] | 2 [1 to 3]
  Severity of wheezing | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 1]
  Severity of numbness/tingling in hands or feet | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 3] | 1.5 [1 to 5] | 1 [1 to 4] | 3 [1 to 3]
  Numbness or tingling in hands or feet interference: number analyzed (Participants) | 17 | 10 | 10 | 10 | 7 | 5
  Numbness or tingling in hands or feet interference | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 4] | 1 [1 to 4] | 3 [1 to 4]
  Severity of dizziness | 1 [1 to 5] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
  Dizziness interference: number analyzed (Participants) | 17 | 10 | 11 | 9 | 6 | 5
  Dizziness interference | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 1] | 1 [1 to 2]
  Severity of concentration problems | 1 [1 to 3] | 1 [1 to 4] | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2]
  Concentration problems interference | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2]
  Severity of memory problems | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1.5 [1 to 3] | 2 [1 to 3] | 1 [1 to 2]
  Memory problem interference: number analyzed (Participants) | 18 | 10 | 11 | 10 | 7 | 5
  Memory problem interference | 1 [1 to 3] | 1.5 [1 to 3] | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2]
  Frequency of pain | 2 [1 to 5] | 3 [1 to 5] | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 5] | 2 [2 to 5]
  Severity of pain | 2 [1 to 5] | 3 [1 to 5] | 2 [1 to 5] | 1.5 [1 to 4] | 2 [1 to 4] | 2 [2 to 3]
  Pain interference: number analyzed (Participants) | 18 | 10 | 11 | 9 | 7 | 5
  Pain interference | 1 [1 to 5] | 3.5 [1 to 5] | 1 [1 to 5] | 1 [1 to 4] | 1 [1 to 4] | 2 [1 to 4]
  Severity of insomnia | 3 [1 to 4] | 2 [1 to 5] | 2 [1 to 3] | 2 [1 to 3] | 3 [1 to 3] | 2 [1 to 3]
  Insomnia interference: number analyzed (Participants) | 18 | 10 | 11 | 10 | 7 | 5
  Insomnia interference | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 3] | 1.5 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
  Severity of fatigue: number analyzed (Participants) | 17 | 11 | 11 | 10 | 7 | 5
  Severity of fatigue | 3 [1 to 5] | 3 [2 to 5] | 3 [2 to 5] | 2.5 [2 to 4] | 3 [2 to 3] | 3 [2 to 3]
  Fatigue interference | 2.5 [1 to 5] | 3 [1 to 5] | 2 [2 to 5] | 2 [1 to 4] | 3 [1 to 3] | 2 [2 to 3]
  Frequency of anxiety | 2 [1 to 4] | 1 [1 to 3] | 2 [1 to 3] | 1.5 [1 to 3] | 1 [1 to 3] | 2 [1 to 2]
  Severity of anxiety | 2 [1 to 4] | 1 [1 to 4] | 2 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 2 [1 to 2]
  Anxiety interference: number analyzed (Participants) | 18 | 11 | 10 | 10 | 7 | 5
  Anxiety interference | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 2]
  Frequency of depression | 1.5 [1 to 3] | 1 [1 to 4] | 1 [1 to 3] | 1.5 [1 to 3] | 1 [1 to 3] | 1 [1 to 3]
  Severity of depression | 1.5 [1 to 3] | 1 [1 to 4] | 1 [1 to 4] | 1.5 [1 to 4] | 1 [1 to 3] | 1 [1 to 3]
  Depression interference: number analyzed (Participants) | 18 | 10 | 11 | 10 | 7 | 5
  Depression interference | 1 [1 to 3] | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2]
  Frequency of sadness or unhappiness: number analyzed (Participants) | 18 | 11 | 9 | 10 | 7 | 5
  Frequency of sadness or unhappiness | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 3] | 2 [1 to 3] | 1 [1 to 3]
  Severity of sadness or unhappiness: number analyzed (Participants) | 18 | 11 | 10 | 10 | 7 | 5
  Severity of sadness or unhappiness | 2 [1 to 3] | 2 [1 to 4] | 1.5 [1 to 4] | 2 [1 to 4] | 2 [1 to 3] | 1 [1 to 2]
  Sadness or happiness interference: number analyzed (Participants) | 18 | 11 | 10 | 10 | 7 | 5
  Sadness or happiness interference | 1 [1 to 3] | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 3] | 1 [1 to 2] | 1 [1 to 2]

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were collected from start of treatment through 360 days following completion of radiotherapy.
Arm/Group | SBRT
All-Cause Mortality (participants affected / at risk) | 33/66
Serious Adverse Events (participants affected / at risk) | 42/66
Other Adverse Events (participants affected / at risk) | 31/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT (N=66)
Abdominal pain (Gastrointestinal disorders) | 3
Accidental morphine overdose (General disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Adenovirus upper respiratory infection (Infections and infestations) | 1
Anal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Blood bilirubin increased (Investigations) | 1
COVID19 (Infections and infestations) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Disease progression (General disorders) | 28
Diverticulitis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Heart failure (Cardiac disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Infection attributed to port (Infections and infestations) | 1
Intracranial hemorrhage (Nervous system disorders) | 2
Jejunal obstruction (Gastrointestinal disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lung infection (Infections and infestations) | 1
Mass on right ventricle (Cardiac disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Post-menopause bleeding (Reproductive system and breast disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1
Stroke (Nervous system disorders) | 1
THA failure with pseudotumor formation (General disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT (N=66)
Abdominal pain (Gastrointestinal disorders) | 8
Acute pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 2
Gastritis (epigastric pain) (Gastrointestinal disorders) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hyponatremia (Investigations) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain (pelvis/hip) (General disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT04553471/Prot_SAP_000.pdf